CLINICAL TRIAL: NCT02021240
Title: Effects of Ketamine in Post-operative Pain and Recovery Outcomes in Bilateral Third Molar Surgery Under General Anaesthesia
Brief Title: Ketamine in Post-operative Dental Pain and Recovery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Wai Cheung, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW13-525
Record Dates: First submitted 2013-12-11; First posted 2013-12-27 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketamine (Active Comparator): Single dose of intravenous ketamine 0.5mg/kg before incision
  Interventions: Drug: Ketamine
- Dexamethasone (Active Comparator): Single dose of intravenous dexamethasone 8mg before incision
  Interventions: Drug: Dexamethasone
- Normal saline (Placebo Comparator): Single dose of intravenous normal saline before incision
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ketamine
  Arms: Ketamine
Drug: Dexamethasone
  Arms: Dexamethasone
Drug: Normal Saline
  Arms: Normal saline

SUMMARY:
Low dose sub-anaesthetic dose of ketamine has been shown to reduce postoperative pain and analgesic consumption. However, due to the heterogeneous results, the standard dosing regimen has not been available. Recently, its effect in postoperative outcomes and the development of post-operative surgical pain has also been suggested.

Ketamine has been shown to reduce post-operative early inflammation especially serum IL-6. Therefore, study in its effects in post- operative pain and outcomes due to inflammation is suggested. Only few clinical studies assessed post-operative pain are related to inflammation.

Pain after third molar surgery is a good model of postoperative acute inflammatory pain.

A previous study showed that there was no benefit to administer ketamine before or after oral surgery for pain relief. However, other studies demonstrated that ketamine used as sedative or local ketamine in third molar surgery could reduce postoperative dental pain, swelling and trismus.

Postsurgical facial oedema is difficult to quantify accurately as it is three dimensional. Over the years, various measurement techniques have been tried to measure oedema objectively. These include direct linear measurement using tape or flexible rulers across fixed soft tissue landmarks, standardized stereophotographic measurements, computerized tomography (CT), magnetic resonance imaging (MRI), ultrasonography (US) and three - dimensional (3D) laser scanning. Recently, three dimensional image reconstructions using a reversed engineering technique has been developed and is used in the manufacturing industry. This technology could be applied in a clinical setting for monitoring soft tissue changes.

In this study, the investigators will aim to study the use of sub-anaesthetic dose of ketamine in post-operative dental pain and recovery outcomes.

The investigators hypothesise that post-operative pain after Bilateral Third Molar under General Anaesthesia is less in patients receiving sub-anaesthetic does of ketamine before incision. The magnitude of this effect will be compared with a positive control group (dexamethasone) as well as a placebo group (normal saline). Further, the investigators aim to demonstrate whether ketamine can reduce post-operative facial oedema and other post-operative outcomes.

DETAILED DESCRIPTION:
3 groups:

Ketamine group:

• Patient will receive single dose of intravenous ketamine 0.5mg/kg before incision.

Dexamethasone group:

* Patient will receive single dose of intravenous dexamethasone 8mg before incision Control group
* Patient will receive single dose of intravenous normal saline before incision.

Process:

After obtaining informed consent, patient will be randomly allocated to one of three groups. HADS and SF-36 questionnaires will be completed by the patients on admission. Blood for serum IL-6 and TNF - α will be taken. 3D laser scanning of the face will be performed.

The patients will not receive any premedication and will follow other routine preoperative preparation. Patients will be educated to use the Numerical Pain Rating Scale for pain assessment, where 0= no pain and 10 the most severe pain. P deletion test and mini-mental test will be done at ward before operation.

Before induction, ketamine 0.5mg/kg, dexamethasone 8mg or normal saline of same volume will be administrated intravenously according to the study group allocated. Induction of anaesthesia will be achieved according to a standard protocol. Regional block with 2% lignocaine with 1 in 80000 adrenaline will be performed by surgeon before start of the procedure. The surgery will be started once the anaesthesia is effective.

The patients will be transferred to the recovery area for monitoring for at least 30 minutes postoperatively. The vital signs including blood pressure, pulse and SpO2 and the Ramsay sedation score (RSS) will be assessed every 5 minutes. Pain score (NRS) will be recorded every 15 minutes. The patients will be sent back to general ward when the parameters are normal. P deletion test will be done from postoperative hour 2 in the general ward until the performance is at least the same as that before operation. Mini-mental test will be done at 2 hours postoperatively. Hourly blood pressure, pulse, SpO2 and pain score (NRS) will be performed for 4 hours. Pain score (NRS) will be assessed 4 hourly afterward. Quality of recovery will be assessed after operation with Chinese QoR. Serum IL-6 and TNF-α will be taken at postoperative 6th hour and 16th hour. Paracetamol 1 g three times daily and tramadol 50mg three times daily as required will be prescribed postoperatively.

The patients will be discharged home at postoperative day 1 if the discharge criteria are met. 3D laser scanning of the face will be performed before they are discharged. They will be asked the degree of satisfaction of the operation . Paracetamol 1 g three times daily and tramadol 50mg three times daily as required will be prescribed on discharge. A diary will be given to the patient. From postoperative day 1 to day 3, at each morning, average pain score (NRS), analgesic consumption and side effects will be marked on the diary by the patient. At the 3rd month after operation, the severity and nature of pain at the surgical sites will be asked over phone. The patients will be asked to go to the Oral & Maxillofacial Surgery out-patient clinic at the Prince Philip Dental Hospital on postoperative day 2 for 3D laser scanning of the face.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* Bilateral wisdom teeth extraction under general anaesthesia
* Age over 18
* Written informed consent

Exclusion Criteria:

* Allergy to ketamine or dexamethasone
* Patient refusal
* Pregnancy
* Alcohol or drug abuse
* Known impaired renal function and liver function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-02-10 (Actual); Primary Completion 2015-09-18 (Actual); Study Completion 2016-04-18 (Actual)

PRIMARY OUTCOMES:
Pain scores as numerical rating scale after operation | Every 15 minutes for 1 hour after operation, every 4 hourly at the first 24 hour after operation, and at postoperative 48th and 72rd hour

SECONDARY OUTCOMES:
Facial oedema measured by using 3D laser scanning of the face | Before operation and at post-operative day1 and day 2
Number of patients having adverse effects | Postoperative day 1 to day 3
Serum IL-6 and TNF - α | Before operation and at postoperative 6th and 16th hour

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wai Cheung, Study Director — Department of Anaesthesiology, Queen Mary Hospital, Hong Kong
Locations (1):
- Oral and Maxillofacial Surgery, Faculty of Dentistry, The University of Hong Kong, Hong Kong, Hong Kong